CLINICAL TRIAL: NCT00047619
Title: Enhancement of Pressure Healing With Pulsatile Lavage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A2803-R
Record Dates: First submitted 2002-10-09; First posted 2002-10-10 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-09

CONDITIONS: Spinal Cord Injury
Keywords: Decubitus Ulcers; Pulsatile Lavage; SCI; Spinal Cord Injury; Wound healing; pressure ulcer
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulsatile lavage group (Experimental): pulsatile lavage therapy
  Interventions: Procedure: Pulsatile Lavage
- Sham lavage group (Sham Comparator): sham pulsatile lavage
  Interventions: Other: sham pulsatile lavage

INTERVENTIONS:
Procedure: Pulsatile Lavage — pulsatile lavage to wound bed
  Arms: Pulsatile lavage group
Other: sham pulsatile lavage — pulsatile lavage to not directed at wound or patient
  Arms: Sham lavage group

SUMMARY:
The purpose of this study is to investigate the use of pulsatile lavage to enhance the healing of pressure ulcers in individuals with spinal cord injury (SCI).

The goals will be achieved using a repeated-measures double-blinded randomized controlled study of individuals with SCI who have pelvic region pressure ulcers. A total of 60 subjects will be recruited to this study. Participants will be randomly assigned to a treatment or control group. Pulsatile lavage treatment will be administered to the treatment group daily for a 3 week period. The control group subjects will receive daily sham pulsatile lavage treatment for 3 weeks. All subjects will be monitored for a 3 week period and will continue to receive routine pressure ulcer care, i.e. dressings and bedrest with a regular turning regime during their participation in the study.

All study participants will be monitored following the study period until complete closure of the pressure ulcer is achieved in order to determine total interval to final closure, including any surgical procedures required. In addition, the economic effects of pulsatile lavage treatment will be evaluated through monitoring of data collected in the Computerized Patient Record System (CPRS), including duration of admission, duration of total bedrest order and duration of treatment for pressure ulcer. This data will give an initial measure of the cost benefits that may be achieved with the use of pulsatile lavage for the treatment of pressure ulcers.

Subjects will be recruited from the Louis Stokes Cleveland Veterans Affairs Medical Center (CVAMC). All individuals with spinal cord injury who are admitted to the SCI Unit with pelvic region pressure ulcers will be considered eligible for this study. Further selection criteria will be employed to screen potential participants as described below. On recruitment subjects will be randomly assigned to 2 groups of 20 subjects. The assessment methods employed will be the same for each volunteer. One group will participate in the pulsatile lavage intervention, the second group will act as controls.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the use of pulsatile lavage to enhance the healing of pressure ulcers in individuals with spinal cord injury (SCI). It will investigate the hypothesis that the treatment of non-necrotic pressure ulcers with pulsatile lavage will enhance the rate of healing.

These goals will be achieved using a repeated-measures double-blinded randomized controlled study of individuals with SCI who have pelvic region pressure ulcers. A total of 60 subjects will be recruited to this study. Participants will be randomly assigned to a treatment or control group. Pulsatile lavage treatment will be administered to the treatment group daily for a 3 week period. The control group subjects will receive daily sham pulsatile lavage treatment for 3 weeks. All subjects will be monitored for a 3 week period and will continue to receive routine pressure ulcer care, i.e. dressings and bedrest with a regular turning regime during their participation in the study.

All study participants will be monitored following the study period until complete closure of the pressure ulcer is achieved in order to determine total interval to final closure, including any surgical procedures required. In addition, the economic effects of pulsatile lavage treatment will be evaluated through monitoring of data collected in CPRS, including duration of admission, duration of total bedrest order and duration of treatment for pressure ulcer. This data will give an initial measure of the cost benefits that may be achieved with the use of pulsatile lavage for the treatment of pressure ulcers.

Methodology Eligible individuals with SCI who are admitted to CVAMC with pelvic region pressure ulcers will be assigned to a pulsatile lavage treatment group or to a second non-intervention control group. A comprehensive assessment methodology will be employed to characterize pressure ulcer healing. All study participants will be assessed at routine intervals using objective measurement techniques. Statistical analysis of inter-group differences will allow the efficacy of pulsatile lavage for pressure ulcer healing to be established. Forty subjects will be enrolled in the study.

Patient Selection Criteria: Subjects will be recruited from the Louis Stokes Cleveland Veterans Affairs Medical Center (CVAMC). All individuals with spinal cord injury who are admitted to the SCI Unit with pelvic region pressure ulcers will be considered eligible for this study. Further selection criteria will be employed to screen potential participants as described below. On recruitment subjects will be randomly assigned to 2 groups of 20 subjects. The assessment methods employed will be the same for each volunteer. One group will participate in the pulsatile lavage intervention, the second group will act as controls.

ELIGIBILITY:
Inclusion Criteria:

Spinal Cord Injury

Exclusion Criteria:

systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2002-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chester H. Ho, MD, Principal Investigator — VA Medical Center-Cleveland
Locations (1):
- VA Medical Center, Cleveland, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Ho CH, Bensitel T, Wang X, Bogie KM. Pulsatile lavage for the enhancement of pressure ulcer healing: a randomized controlled trial. Phys Ther. 2012 Jan;92(1):38-48. doi: 10.2522/ptj.20100349. Epub 2011 Sep 23. PMID 21949432

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulsatile Lavage Group | Sham Lavage Group
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham Lavage Group: sham pulsatile lavage
  sham pulsatile lavage: pulsatile lavage not directed at wound or patient
- Total: Total of all reporting groups
Arm/Group | Pulsatile Lavage Group | Sham Lavage Group | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Customized [Number; unit: participants] — Age above 18 who can give appropriate consent to the study
  participants
    Number of subjects >=18 years | 14 | 14 | 28
Sex/Gender, Customized [Number; unit: participants] — Both male and female subjects are eligible, though recruitment in the veterans affairs medical center spinal cord injury service resulted in only males being recruited as there were very few females with spinal cord injury in the veterans affairs medical center spinal cord injury service.
  participants
    male gender | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Pressure Ulcer Geometry
Description: Linear assessment of wounds
Time Frame: study participation - up to 6 weeks
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Pulsatile Lavage Group | Sham Lavage Group
Number analyzed (Participants) | 14 | 14
cm
  Length in cm | 3.5 [2.47 to 4.54] | 4.9 [3.53 to 6.32]
  Width in cm | 2.9 [1.92 to 3.78] | 3.0 [1.30 to 4.65]
  Depth in cm | 1.4 [0.59 to 2.20] | 2.5 [1.81 to 3.16]

2. Primary Outcome: Pressure Ulcer Volume Measurement
Description: Volume of pressure ulcer was measured by the amount of fluid that could be used to fill the pressure ulcer which was covered by an occlusive dressing
Time Frame: study participation - up to 6 weeks
Measure: Mean (95% Confidence Interval); unit: cm^3
Arm/Group | Pulsatile Lavage Group | Sham Lavage Group
Number analyzed (Participants) | 14 | 14
cm^3 | 5.8 [2.79 to 8.79] | 12.4 [8.39 to 16.38]

ADVERSE EVENTS:
Time Frame: Duration of study
Arm/Group | Pulsatile Lavage Group | Sham Lavage Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No